CLINICAL TRIAL: NCT05229926
Title: Implementation of CareCube Negative Pressure Isolation Units in a High-Volume Tertiary Care Hospital: A Pilot Study
Brief Title: Implementation of CareCube Negative Pressure Isolation Units
Acronym: CareCube
Status: Completed | Type: Observational
Sponsor: Saint Luke's Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 21-024
Record Dates: First submitted 2021-10-12; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Infectious Disease
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient Group: Patients who previously were hospitalized during the COVID-19 pandemic, receiving mock care inside the CareCube
  Interventions: Device: CareCube
- Patient Caregiver Group: Caregivers/family/friends of patients previously hospitalized during the COVID-19 pandemic, communicating with the patient inside the CareCube
- Heathcare Provider Group: Physicians, Certified Registered Nurse Anesthetists, RNs, Certified Nursing Assistants who will perform routine clinical care tasks, including passing food and medicines, drawing blood, inserting an IV. To simulate intubation, a mannequin will be used.

INTERVENTIONS:
Device: CareCube — modular, disposable, negative pressure, isolation patient care system
  Groups: Patient Group

SUMMARY:
Pilot study to provide a descriptive analysis of the real-world feasibility of using a CareCube for COVID-19 patients in a high-volume tertiary care hospital.

DETAILED DESCRIPTION:
The CareCube is a modular, disposable, negative pressure, isolation patient care system that can rapidly augment hospital's capacity to care for patients with contagious droplets or airborne pathogens. It is designed as a temporary single-use negative pressure isolation care unit with PPE for common patient care protocols built into the unit. The device is intended to be used in a healthcare setting as a temporary isolation of patients with suspected or confirmed diagnosis of COVID-19 to prevent Healthcare Practitioners (HCP) and patients' visitors from being exposed to pathogenic biological airborne particulates. The system includes three components: an isolation chamber, functional gown, and gloves. The isolation chamber functions in a similar manner to a hospital negative pressure, Airborne Infection Isolation Room. The gown and gloves provide an extra layer of barrier protection beyond PPE. The CareCube is designed to provide improved protection for front-line healthcare workers, while also conserving the vital supplies of N95 masks, face shields, and gowns, which are not required since there is no direct contact with the patient.

The goal of this project is to provide preliminary data to describe the experiences of 'patients', their caregivers, and providers with the CareCube.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female previously hospitalized during the COVID-19 pandemic
* At least 21 days post- positive COVID-19 test result
* Able to provide written informed consent

Exclusion Criteria:

* Under 18 years of age
* Unable to provide written informed consent on own behalf

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eight patients who previously were hospitalized during the COVID-19 pandemic, were approached for participation, along with their caregivers (family, friend or home nurse, who would regularly visit the patient in the hospital), if applicable. Patients were at least 21 days removed from a positive COVD-19 test, thus meeting and exceeding CDC guidelines for post COVID quarantine. Six healthcare providers (doctors, CRNAs, RNs, CNAs) were also recruited.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-03-27 (Actual); Primary Completion 2021-03-27 (Actual); Study Completion 2021-03-27 (Actual)

PRIMARY OUTCOMES:
Completion of Nursing Assistant Task - Nasal Swab | through study completion, one day
  success of obtaining nasal swab as assessed by observer (successful/not successful)
Completion of Nursing Assistant Task - Obtain Patient Weight | through study completion, one day
  success of obtaining patient weight as assessed by observer (successful/not successful)
Completion of Nursing Assistant Task - Obtain Vital Signs | through study completion, one day
  success of obtaining vital signs as assessed by observer (successful/not successful)
Completion of Nursing Assistant Task - Attach Telemetry Stickers | through study completion, one day
  success of telemetry stickers attachment as assessed by observer (successful/not successful)
Completion of Nursing Assistant Task - Place Nasal Cannula | through study completion, one day
  success of nasal cannula O2 placement as assessed by observer (successful/not successful)
Completion of Nursing Assistant Task - Pass Through Tray | through study completion, one day
  success of passing a tray of food via pass-through to patient as assessed by observer (successful/not successful)
Completion of Nursing Assistant Task - Receive Tray | through study completion, one day
  success of collecting a tray of food/waste/ via pass-through from the patient as assessed by observer (successful/not successful)
Completion of Registered Nurse Task - Medications | through study completion, one day
  success of medicine reconciliation (generic medication questions, i.e., do you take an aspirin, etc.) with patient as assessed by observer (successful/not successful)
Completion of Registered Nurse Task - Place Nasal Cannula | through study completion, one day
  success of nasal cannula O2 placement as assessed by observer (successful/not successful)
Completion of Registered Nurse Task - Place Non-Rebreather Mask | through study completion, one day
  success of non-rebreather mask placement as assessed by observer (successful/not successful)
Completion of Registered Nurse Task - Place Intravenous Line | through study completion, one day
  success of intravenous line placement as assessed by observer (successful/not successful)
Completion of CRNA Task (Mannequin) - Intubation | through study completion, one day
  success of intubation as assessed by observer (successful/not successful)
Completion of CRNA Task (Mannequin) - Attach Defibrillator Pads | through study completion, one day
  success of external defibrillator pad placement as assessed by observer (successful/not successful)

SECONDARY OUTCOMES:
Caregiver Satisfaction | through study completion, one day
  level of satisfaction based on completion of caregiver survey
Healthcare Provider Satisfaction | through study completion, one day
  level of satisfaction based on completion of provider survey
Patient Experience of Claustrophobia | through study completion, one day
  subject experience based on claustrophobia assessment
Patient Experience of Stress and Anxiety | through study completion, one day
  subject experience based on completion of STAIAD
Patient Satisfaction | through study completion, one day
  level of satisfaction based on completion of patient survey

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Luke's Hospital of Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data

REFERENCES:
- [Background] Jones DS. History in a Crisis - Lessons for Covid-19. N Engl J Med. 2020 Apr 30;382(18):1681-1683. doi: 10.1056/NEJMp2004361. Epub 2020 Mar 12. No abstract available. PMID 32163699
- [Background] Ortega R, Gonzalez M, Nozari A, Canelli R. Personal Protective Equipment and Covid-19. N Engl J Med. 2020 Jun 25;382(26):e105. doi: 10.1056/NEJMvcm2014809. Epub 2020 May 19. No abstract available. PMID 32427435
- [Background] Al-Benna S. Negative pressure rooms and COVID-19. J Perioper Pract. 2021 Jan-Feb;31(1-2):18-23. doi: 10.1177/1750458920949453. Epub 2020 Dec 1. PMID 33353524
- [Background] Winck JC, Ambrosino N. COVID-19 pandemic and non invasive respiratory management: Every Goliath needs a David. An evidence based evaluation of problems. Pulmonology. 2020 Jul-Aug;26(4):213-220. doi: 10.1016/j.pulmoe.2020.04.013. Epub 2020 Apr 27. PMID 32362507
- [Background] Lenaghan PA, Schwedhelm M. Nebraska biocontainment unit design and operations. J Nurs Adm. 2015 Jun;45(6):298-301. doi: 10.1097/NNA.0000000000000202. PMID 26010276
- [Background] Spielberger C, Gorsuch R, Lushene R, Vagg PR and Jacobs G. Manual for the State-Trait Anxiety Inventory (Form Y1 - Y2); 1983.
- [Background] Vujanovic AA, Arrindell WA, Bernstein A, Norton PJ, Zvolensky MJ. Sixteen-item Anxiety Sensitivity Index: confirmatory factor analytic evidence, internal consistency, and construct validity in a young adult sample from the Netherlands. Assessment. 2007 Jun;14(2):129-43. doi: 10.1177/1073191106295053. PMID 17504886
- [Background] Pull CB. [DSM-IV]. Encephale. 1995 Dec;21 Spec No 5:15-20. French. PMID 8582301